CLINICAL TRIAL: NCT01769950
Title: Evaluation of the Incidence of Choline-PET Detected Nodal Metastases Among Newly Diagnosed Prostate Cancer Patients With Presumed Absence of Nodal and Distant Metastases.
Brief Title: Choline-PET for Evaluating the Incidence of Nodal Metastases Among Newly Diagnosed Patients of Prostate Cancer
Acronym: ChoPEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangalore Institute of Oncology (Other)
Responsible Party: Principal Investigator, Sridhar P Susheela, Principal Investigator, Bangalore Institute of Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Choline-Prostate-1
Record Dates: First submitted 2013-01-10; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Choline PET; Choline PET-CT; Positron emission tomography; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Choline-PET arm (Experimental): Every eligible patient will be scanned with Choline-PET at the time of diagnosis of prostate cancer. MRI will also be obtained as it is the current standard of care. CT scan will be obtained as part of the same procedure while procuring the Choline-PET scan with PET-CT dual imaging hardware.
  Interventions: Other: Choline-PET

INTERVENTIONS:
Other: Choline-PET — Carbon-11 or Fluorine-18 PET-CT will be acquired with a scanner with integrated PET and CT scanning ability at the time of diagnosis. It must be however noted that Choline-PET will not be considered as an alternative to magnetic resonance imaging (MRI). In fact, all patients will undergo MRI too.
  Other Names: Choline PET-CT; Choline PET/CT; Carbon-11 Choline PET; Fluorine-18 Choline PET

SUMMARY:
Nodal involvement among patients with prostate cancer is known to be a poor prognostic factor. Traditionally, the presence or absence of nodal disease in patients with prostate cancer is ascertained with the use of anatomical imaging methods such as computed tomography (CT) and magnetic resonance imaging (MRI).

However, the sensitivities of CT and MRI for the detection of pelvic nodal disease is rather low, with reports placing the value to lie between 50-80%.

Positron emission tomography (PET) with the use of carbon-11 or fluorine-18 tagged choline (Choline-PET) is an approach which is known to deliver a high sensitivity for the imaging of prostate cancer disease burden in the primary, nodal and the metastatic areas.

The investigators in this prospective trial intend to utilize Choline-PET among all newly diagnosed patients of prostate cancer who are presumed to be non-N1 (absence of nodal disease on conventional imaging) and non-M1 (absence of metastatic disease on conventional imaging).

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients
* Diagnosed prostate cancer

Exclusion Criteria:

* Metastatic disease at presentation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Detection of Choline-PET detected nodal metastases | Eligible participants will undergo a Choline-PET scan before the initiation of any cancer specific treatments, that is within a time frame of one week from the time of diagnosis
  At the time of diagnosis of prostate cancer, the investigators intend to utilize Choline-PET scan to gain evidence of nodal metastatic disease with a motive to assess for a potentially higher sensitivity than with the use of conventional imaging methods such as CT or MRI.

SECONDARY OUTCOMES:
Comparison of Choline-PET and CT for the detection of nodal metastatic disease | Eligible participants will undergo a Choline-PET scan before the initiation of any cancer specific treatments, that is within a time frame of one week from the time of diagnosis
  For each enrolled patient, the information regarding nodal metastatic disease gained from Choline-PET scan will be compared with CT scan data.
Comparison of Choline-PET and MRI for the detection of nodal metastatic disease | Eligible participants will undergo a Choline-PET scan before the initiation of any cancer specific treatments, that is within a time frame of one week from the time of diagnosis
  For each enrolled patient, the information regarding nodal metastatic disease gained from Choline-PET scan will be compared with MRI scan data.

OTHER OUTCOMES:
Detection of extra-pelvic non-nodal metastases | Eligible participants will undergo a Choline-PET scan before the initiation of any cancer specific treatments, that is within a time frame of one week from the time of diagnosis
  Evidence of extra-pelvic non-nodal metastases detected by Choline-PET scan will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ajaikumar Basavalingaiah, MD, Study Chair — HealthCare Global- Bangalore Insititute of Oncology; Kumar G Kallur, MD, Study Director — HealthCare Global- Bangalore Institute of Oncology; Swaroop Revannasiddaiah, MD, Study Director — HealthCare Global- Bangalore Institute of Oncology; Sandeep Muzumder, MD, Study Director — HealthCare Global- Bangalore Institute of Oncology; Govindarajan Mallarajapatna, MD, Study Director — HealthCare Global- Bangalore Institute of Oncology; Raghunath S Krishnappa, MS, DNB, Study Director — HealthCare Global- Bangalore Institute of Oncology
Locations (1):
- HealthCare Global- Bangalore Institute of Oncology, Bengaluru, Karnataka, India